CLINICAL TRIAL: NCT04933214
Title: Adherence to Exclusive Enteral Nutrition in Patients With Crohn's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0324
Record Dates: First submitted 2021-06-17; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-05

CONDITIONS: Crohn Disease
Keywords: Crohn's disease, Exclusive Enteral Nutrition, Adherence
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study has not yet been completed

ELIGIBILITY:
Inclusion Criteria:

* The main inclusion criteria were as follows: had diagnosed CD more than 3 months; had EEN in the past 6 months; were at least 18 years old; agreed to participate in this study.

Exclusion Criteria:

* The exclusion criteria were received treatment from mental health professionals due to any mental or cognitive impairment; suffered from other serious diseases, such as heart, brain, lung, liver and kidney dysfunction; severe infection, anemia, cachexia or other serious complications were found.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We investigated CD patients who received EEN therapy in tertiary hospital in Hangzhou from December 2020 to May 2021.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Estimated)
Dates: Start 2021-05-12 (Actual); Primary Completion 2021-12-12 (Estimated); Study Completion 2021-12-12 (Estimated)

PRIMARY OUTCOMES:
Adherence | December 2020 to May 2021
  The adherence of patients was evaluated by the ratio of daily actual intake of energy to daily target energy.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Chen, Study Director — 2ndAffiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2ndAffiliated Hospital, School of Medicine, Zhejiang University, China, Zhejiang, China